CLINICAL TRIAL: NCT04911413
Title: Comparison of Three Tranexamic Acid Dose Regimens in Patients Undergoing Cardiac Valve Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, SHI Jia, Director，the department of Anesthesiology, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TXA dosage trial 2
Record Dates: First submitted 2021-05-25; First posted 2021-06-03 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Cardiac Surgical Procedures; Blood Transfusion; Tranexamic Acid
Keywords: Cardiac Surgery; Blood transfusion; Blood loss; Tranexamic Acid; Dose regimen
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low-dose group, (Experimental): A bolus of 10 mg/kg Tranexamic Acid followed by a maintenance dose of 10 mg/kg/h Tranexamic Acid until the end of surgery
  Interventions: Drug: Tranexamic acid
- middle-dose group, (Experimental): A bolus of 20 mg/kg Tranexamic Acid followed by a maintenance dose of 15 mg/kg/h Tranexamic Acid until the end of surgery
  Interventions: Drug: Tranexamic acid
- high-dose group (Experimental): A bolus of 30 mg/kg Tranexamic Acid followed by a maintenance dose of 20 mg/kg/h Tranexamic Acid until the end of surgery
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — The drug used in this RCT is tranexamic acid. We used three different doses of TXA in three groups.
  Other Names: Cyklokapron; Transamin

SUMMARY:
This study compares the effect of three different dose levels of tranexamic acid（TXA）in reducing blood loss and transfusion requirements in cardiac valve surgery.

DETAILED DESCRIPTION:
The effect of TXA to reduce perioperative blood loss and blood transfusion has been well established in many trials, but the optimal dosage of TXA in cardiac surgery has always been a problem of debate. This is a single-center randomized controlled trial to study different dose regimens of TXA in cardiac surgery. We use three different dose levels of TXA in cardiac valve surgery with CPB, and see if there are any differences in perioperative blood loss and transfusion requirements. Serious adverse events and seizure attacks are also recorded until three months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 to 60 years old scheduled for cardiac valve surgery (replacement or plasty) requiring CPB

Exclusion Criteria:

* known allergy to TXA, combined CABG operation or other cardiac procedures other than valve surgery, previous cardiac surgery, EF<45% or cardiothoracic ratio>0.65, serious coagulation disorder, serious hepatic insufficiency, receiving antiplatelet therapy at any time within 7 days of surgery, receiving low molecular weight heparin at any time within 24 hours of surgery, and pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
total postoperative drainage | from the operation day to the discharge，an average of 7 days
  The total chest tube drainage postoperatively

SECONDARY OUTCOMES:
Red blood cells transfusion rate（%），Red blood cells transfusion volume（ml） | from the operation day to the discharge，an average of 7 days
  intraoperative and postoperative RBC transfusion rate and transfusion volume（for all patients and for transfused patients）
Fresh frozen plasma transfusion rate（%），Fresh frozen plasma transfusion volume（ml） | from the operation day to the discharge，an average of 7 days
  intraoperative and postoperative FFP transfusion rate and transfusion volume（for all patients and for transfused patients）
Platelet transfusion rate（%），Platelet transfusion volume（ml） | from the operation day to the discharge，an average of 7 days
  intraoperative and postoperative platelet transfusion rate and transfusion volume（for all patients and for transfused patients）
repeat surgery because of bleeding | from the operation day to the discharge，an average of 7 days
  rate of repeat surgery due to massive bleeding
rate of death | from the operation day to three months after surgery
  rate of death
seizure attack | from the operation day to three months after surgery
  any seizure attack is recorded
length of stay in ICU and hospital | from the operation day to the discharge，an average of 7 days
  the length of stay in ICU and hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No